CLINICAL TRIAL: NCT06356701
Title: A Single-center, Randomized, Controlled Clinical Study Comparing the Efficacy and Safety of Tumor Nutritional Therapy Combined With Immune Checkpoint Inhibitors and Chemotherapy in the First-line Treatment of Stage IV NSCLC Without Driver Gene Mutations
Brief Title: Tumor Nutritional Therapy in the First-line Treatment of Stage IV NSCLC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: dongyandl
Record Dates: First submitted 2024-03-20; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-01

CONDITIONS: Long-Term Effects Secondary to Cancer Therapy
Keywords: lung cancer; Effect of nutritional therapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Cancer nutritional treatment regimen (Spirulina Bifidobacterium Capsules, Fish Oil Grape Seed Blueberry Soft Capsules, Ganoderma Spore Oil Soft Capsules) — Medication for Research :
  * Spirulina Bifidobacterium Capsules
  * Fish Oil Grape Seed Blueberry Soft Capsules;
  * Ganoderma Lucidum Sporoderm Oil Soft Capsules; oral administration. non-squamous cell carcinoma Drug: Pemetrexed+Cisplatin (or carboplatin)
    * Sintilimab Injection/Camrelizumab/Tislelizumab/Atezolizumab Injection IV infusion squamous cell carcinoma Drug:Paclitaxel+ Cisplatin (or carboplatin)
    * Sintilimab Injection/Camrelizumab/Tislelizumab/Atezolizumab Injection IV infusion

SUMMARY:
A Single-center, Randomized, Controlled Clinical Study Comparing the Efficacy and Safety of Tumor Nutritional Therapy Combined With Immune Checkpoint Inhibitors and Chemotherapy in the First-line Treatment of Stage IV NSCLC Without Driver Gene Mutations

DETAILED DESCRIPTION:
Main purpose: Cancer nutritional treatment regimen (Spirulina Bifidobacterium Capsules, Fish Oil Grape Seed Blueberry Soft Capsules, Ganoderma Spore Oil Soft Capsules) combined with immune checkpoint inhibitors and chemotherapy in the first-line treatment of stage IV non-small cell lung cancer without driver gene mutations efficacy in.Secondary purpose: Cancer nutritional treatment regimen (Spirulina Bifidobacterium Capsules, Fish Oil Grape Seed Blueberry Soft Capsules, Ganoderma Spore Oil Soft Capsules) combined with immune checkpoint inhibitors and chemotherapy in the first line of stage IV non-small cell lung cancer without driver gene mutations Safety in treatment.Exploratory purpose: Tumor nutritional treatment regimen (Spirulina Bifidobacterium Capsules, Fish Oil Grape Seed Blueberry Soft Capsules, Ganoderma Spore Oil Soft Capsules) combined with immune checkpoint inhibitors and chemotherapy in the first line of stage IV non-small cell lung cancer without driver gene mutations The relationship between the number of T cell subpopulations and changes in inflammatory factors during treatment and the therapeutic effect, and whether the T cell subpopulation analysis method can effectively monitor and evaluate the status of the tumor immune microenvironment.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in this clinical study
* Fully understand and know this research and sign the informed consent form.
* Be 18-75 years old (inclusive) on the day of signing ICF.
* Stage IV non-small cell lung cancer first diagnosed by histology or cytology. There is no known epidermal growth factor receptor (EGFR) sensitive mutation, anaplasticlymphomakinase (ALK) gene rearrangement and ros sarcoma oncogenic factor 1- receptor tyrosine kinase (ROS1) gene fusion.
* The physical condition of 4.ECOG is 0-2, and the expected survival time is more than three months
* It must have measurable target lesions judged by researchers according to RECIST v1.1.
* Subjects should provide tumor tissue samples collected at or after the diagnosis of stage IV NSCLC, which are fixed by formalin and can be used to determine the expression level of PD-L1.
* Subjects must have sufficient organ function, which is evaluated according to the following laboratory examination results (and have not received medical support treatment such as blood transfusion, infusion of apheresis components, erythropoietin and granulocyte colony stimulating factor within 14 days before the administration of the study drug):
* Except for hearing loss, alopecia and fatigue, all toxicity caused by previous anti-tumor treatments must have been restored to ≤ 1 grade.
* Fertile women must have a serum pregnancy test within 7 days before the first medication, and the result is negative.
* No obvious heart disease, no myocardial infarction in the past 6 months. Obvious congestive heart failure, obvious supraventricular arrhythmia, conduction block above grade II, acute myocardial ischemia or prolonged QT interval.
* No antibiotics, probiotic foods or microecological agents were used in the first two weeks.

Exclusion Criteria:

* Histologically identified as small cell lung cancer or with small cell components
* Active or untreated central nervous system metastasis and/or cancerous meningitis.
* Received major surgery except diagnostic biopsy within 4 weeks before the first medication, and received radical radiotherapy within 6 months before medication.
* People with active autoimmune diseases, or those who have suffered from autoimmune diseases and are likely to recur.
* Currently receiving systemic hormone therapy or using any other form of immunosuppressive therapy within 14 days before the first administration.
* Other primary malignant tumors have appeared in the past five years, except for locally curable malignant tumors after radical treatment.
* Have received any antibody/drug (including PD-1, PD-L1, CTLA4, TIM3, LAG3, etc.) targeting T cell co-regulatory proteins (immune checkpoints).
* Suffering from interstitial lung disease, or having a history of interstitial lung disease in the past and needing hormone therapy
* Previous history of idiopathic pulmonary fibrosis, drug-induced pneumonia, organized pneumonia and idiopathic pneumonia
* Or those with active pneumonia proved by chest CT in screening period.
* Received live vaccine inoculation within 28 days before the first drug administration.
* Participated in other clinical research trials within 28 days before the first administration of the research drug, and received research drug treatment or used research equipment.
* Chinese medicines with anti-tumor indications have been used within 14 days before the first administration of the study drug.
* Have a history of inflammatory enteritis or have inflammatory bowel disease (such as Crohn's disease and ulcerative colitis).
* There are serious acute and chronic infections.
* Pleural effusion or pericardial effusion that cannot be controlled after appropriate intervention, or ascites that needs repeated drainage (once a month or more frequently).
* Known history of alcoholism or drug abuse.
* Pregnant or lactating women.
* Have a history of drug allergy, such as pemetrexed, carboplatin, carboplatin or other platinum compounds, or their preventive drugs
* Have an allergic history to paclitaxel or protein-bound paclitaxel components
* Or asthma is not controlled.
* Suffering from major cardiovascular diseases
* Acute myocardial infarction, unstable angina pectoris, stroke and transient ischemic attack occurred in the first 6 months
* Suffering from congestive heart failure (NYHA≥2)
* Severe arrhythmia requiring medical treatment.
* The researcher thinks that the subject's complications or other circumstances may affect the compliance with the protocol or be unsuitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | through study completion, an average of 1 year
  The time from the date of randomization until progression of disease according to RECIST 1.1 and iRECIST or death
Assessment of global disorders in patients with cancer | "through study completion, an average of 1 year".
  Quality of life of patients with NSCLC assessed by QLQ-C30
ORR | through study completion, an average of 1 year
  The percentage of the participants who have a Complete Response or a Partial Response as assessed by a blind independent central reviewer per RECIST 1.1 and iRECIST

CONTACTS AND LOCATIONS:
Locations (1):
- DongYan, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No